CLINICAL TRIAL: NCT05621239
Title: Safety Profile of BNT162b2 mRNA SARS-Cov-2 Vaccine in Indonesia: A National Passive Surveillance.
Brief Title: A Study to Understand is the COVID-19 Vaccine BNT162b2 is Safe in Indonesia People
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591050; NCT05621239 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-11-16; First posted 2022-11-17 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: Indonesia; Vaccine; BNT162b2
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Observational study for secondary data collection and analysis of structured data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COMIRNATY: COVID-19 mRNA vaccine
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — BNT162b2 half dose and full dose

SUMMARY:
The purpose of this study is to characterize descriptively the BNT162b2 vaccination safety experience among the Indonesian people. We will look at adverse events (AEs) reported in Indonesia Vaccine Safety Website for people 12 years of age and older. AEs are unwanted reactions associated with the use of the BNT162b2 vaccine. They may or may not be caused by this vaccine.

The secondary data collection will be exclusively from the Indonesia Vaccine Safety Website as requested by BPOM. This study does not seek additional participants. We will look at reported AEs for BNT162b2 vaccine since it became available in Indonesia. Individual data will be de-identified first before use. This will help protect personal information.

We will study the AEs associated with the BNT162b2 vaccine in several ways. These include the type of AEs and which body parts affected, among others. This will help us understand it the vaccine is safe in Indonesian people.

ELIGIBILITY:
Inclusion Criteria:

This study will include adverse events reported in Indonesia Vaccine Safety Website for individuals 12 years of age and older

Exclusion Criteria:

None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: people in Indonesia above 12 years of age who received vaccine and report an adverse event
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants who received BNT162b2 messenger ribonucleic acid (mRNA) Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2) vaccine and reported adverse events (AE) in Indonesia were analysed in this study.
Pre-assignment Details: This retrospective observational study used data from Indonesia Vaccine Safety Website as requested by Indonesia Food and Drug Monitoring Agency(BPOM). A total of 72,394,389 participants (48,425,165 [primary dose] and 23,969,029 [booster dose] received BNT162b2 mRNA SARS-CoV-2 vaccine. Adverse events were reported in 260 participants following administration of the BNT162b2 mRNA vaccine, starting from the time of vaccine availability in Indonesia and data was obtained for these 260 participants.
Groups:
- BNT162b2 mRNA SARS-CoV-2 Vaccine: Participants vaccinated with BNT162b2 mRNA SARS-CoV-2 vaccine and reported AEs were included in this retrospective observational study.
Period: Overall Study
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Started | 260
Completed | 260
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Number analyzed (Participants) | 260
Age, Customized [Count of Participants; unit: Participants]
  12-17 years | 37
  18-30 years | 78
  31-45 years | 83
  46-59 years | 37
  Greater than (>) 59 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) After Primary Dose
Description: An SAE was any untoward medical occurrence at any dose that: suspected to cause death; required hospitalization; life-threatening; persistent or significant disability/incapacity. The number of participants with SAEs after administration of BNT162b2 mRNA SARS-CoV-2 vaccine primary dose are reported in this outcome measure.
Time Frame: The secondary data analysis of structured AE data conducted from 15-Mar-2023 to 03-Apr-2023(approximately 20 days) included AEs reported following administration of BNT162b2 mRNA SARS-CoV-2 vaccine from 21-Aug-2021 to 14-Dec-2022(approximately 1.3 years)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Groups:
- BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose: Participants vaccinated with primary dose of BNT162b2 mRNA SARS-CoV-2 vaccine and reported AEs were included in this retrospective observational study.
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose
Number analyzed (Participants) | 150
Participants | 16

2. Primary Outcome: Number of Participants With SAEs After Booster Dose
Description: An SAE was any untoward medical occurrence at any dose that: suspected to cause death; required hospitalization; life-threatening; persistent or significant disability/incapacity. The number of participants with SAEs after administration of BNT162b2 mRNA SARS-CoV-2 vaccine booster dose are reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Groups:
- BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose: Participants vaccinated with booster dose of BNT162b2 mRNA SARS-CoV-2 vaccine reporting AEs were included in this retrospective observational study.
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose
Number analyzed (Participants) | 110
Participants | 5

3. Primary Outcome: Number of Participants With Non Serious Adverse Events (Non SAEs) After Primary Dose
Description: An AE was any untoward medical occurrence in a participant; the event need not necessarily have a causal relationship with the treatment. AEs other than SAEs were considered non-SAEs. The number of participants with AEs after administration of BNT162b2 mRNA SARS-CoV-2 vaccine primary dose are reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose
Number analyzed (Participants) | 150
Participants | 134

4. Primary Outcome: Number of Participants With Non SAEs After Booster Dose
Description: An AE was any untoward medical occurrence in a participant; the event need not necessarily have a causal relationship with the treatment. AEs other than SAEs were considered non-SAEs. The number of participants with AEs after administration of BNT162b2 mRNA SARS-CoV-2 vaccine booster dose are reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose
Number analyzed (Participants) | 110
Participants | 105

5. Secondary Outcome: Number of SAEs Reported According to Time of Onset
Description: An SAE was any untoward medical occurrence at any dose that: suspected to cause death; required hospitalization; life-threatening; persistent or significant disability/incapacity. The number of SAEs reported according to time of onset less than equal to (<=30) minutes (min) and more than (>) 30 minutes after administration of BNT162b2 mRNA vaccine primary and booster dose are reported in this outcome measure.
Time Frame: Within 30min and>30min after vacc., secondary data analysis of structured AE data conducted from 15-Mar-2023 to 03-Apr-2023(approximately 20 days)included AEs reported following administration vacc. from 21-Aug-2021 to 14-Dec-2022(approximately 1.3 years)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study. Here " Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Number; unit: Events
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose
Number analyzed (Participants) | 16 | 5
Events
  Onset Interval >30 Mins: Fever | 7 | 3
  Onset Interval >30 Mins: Malaise/Fatigue | 5 | 2
  Onset Interval >30 Mins: Nausea/vomiting | 5 | 2
  Onset Interval >30 Mins: Headache | 3 | 2
  Onset Interval >30 Mins: Local pain | 2 | 1
  Onset Interval >30 Mins: Diarrhea | 3 | 0
  Onset Interval >30 Mins: Arthralgia/myalgia | 1 | 1
  Onset Interval >30 Mins: Chills | 2 | 0
  Onset Interval >30 Mins: Local swelling | 0 | 1
  Onset Interval >30 Mins: Syncope/loss of consciousness | 6 | 1
  Onset Interval >30 Mins: Dyspnea/tachypnea | 3 | 2
  Onset Interval >30 Mins: Stomachache/dyspepsia | 3 | 1
  Onset Interval >30 Mins: Vertigo/dizziness | 4 | 0
  Onset Interval >30 Mins: Seizure | 2 | 1
  Onset Interval >30 Mins: Paralysis/paresis | 2 | 1
  Onset Interval >30 Mins: Slurred speech | 3 | 0
  Onset Interval >30 Mins: Chest pain/chess tightness | 1 | 0
  Onset Interval >30 Mins: Hyperhidrosis | 1 | 0
  Onset Interval >30 Mins: Hypesthesia/paresthesia | 0 | 1
  Onset Interval >30 Mins: Insomnia | 1 | 0
  Onset Interval <=30 Mins: Fatigue | 0 | 1
  Onset Interval <=30 Mins: Syncope | 3 | 0
  Onset Interval <=30 Mins: Dizziness | 0 | 1
  Onset Interval <=30 Mins: Chest pain | 1 | 0
  Onset Interval <=30 Mins: Hyperhidrosis | 0 | 1

6. Secondary Outcome: Number of Participants According to Causality of SAEs
Description: An SAE was any untoward medical occurrence at any dose that: suspected to cause death; required hospitalization; life-threatening; persistent or significant disability/incapacity. The causality of SAEs were classified as coincidence: inconsistent causal association to immunization; vaccine reaction, indeterminate: when adequate information is available but it is not possible to assign it, unclassifiable.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose
Number analyzed (Participants) | 16 | 5
Participants
  Coincidence | 12 | 3
  Vaccine Reaction | 0 | 1
  Unclassifiable | 2 | 0
  Indeterminate | 2 | 1

7. Secondary Outcome: Number of Participants According to Type of AEs
Description: AEs can be categorised into SAEs and non-SAEs. SAE was any untoward medical occurrence at any dose that: suspected to cause death; required hospitalization; life-threatening; persistent or significant disability/incapacity. An AE was any untoward medical occurrence in a participant; the event need not necessarily have a causal relationship with the treatment. AEs other than SAEs were considered non-SAEs.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Number analyzed (Participants) | 260
Participants
  SAEs | 21
  Non SAEs | 239

8. Secondary Outcome: Number of AEs Reported According to Solicited and Unsolicited AEs
Description: An AE was any untoward medical occurrence in a participant; the event need not necessarily have a causal relationship with the treatment. Solicited AEs are reported and are part of the uniform collection of information in the registry and unsolicited AEs are volunteered or noted in an unsolicited manner and not as a required data element through a case report form.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Events
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Number analyzed (Participants) | 260
Events
  Solicited | 359
  Unsolicited | 154

9. Secondary Outcome: Number and Type of Solicited AEs Reported
Description: An AE was any untoward medical occurrence in a participant who received BNT162b2 mRNA SARS-CoV-2 vaccine; the event need not necessarily have a causal relationship with the treatment. Solicited AEs are reported and are part of the uniform collection of information in the registry. These were classified as local reactions (local pain, local swelling, local erythema) and systemic reactions (fever, nausea/vomitus, headache, malaise/fatigue, arthralgia/myalgia, chill and diarrhea).
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Events
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Number analyzed (Participants) | 260
Events
  Local pain | 48
  Local swelling | 24
  Local erythema | 7
  Fever | 113
  Nausea/vomiting | 51
  Headache | 43
  Malaise/fatigue | 34
  Arthralgia/myalgia | 17
  Chills | 11
  Diarrhea | 11

10. Secondary Outcome: Number and Type of Unsolicited AEs Reported
Description: An AE was any untoward medical occurrence in a participant who received BNT162b2 mRNA SARS-CoV-2 vaccine; the event need not necessarily have a causal relationship with the treatment. Unsolicited AEs are volunteered or noted in an unsolicited manner and not as a required data element through a case report form. These were classified as local reactions (local sore, local itch and erythema) and systemic reactions (vertigo/dizziness, cough/rhinitis/sore throat, itchy, dyspnea/tachypnea, drowsiness, syncope/loss of consciousness, hypesthesia/paresthesia, chest pain/chest tightness, stomach ache/dyspepsia, seizure, paralysis/paresis, slurred speech, hyperhidrosis and insomnia).
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Number; unit: Events
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine
Number analyzed (Participants) | 260
Events
  Local sore | 10
  Local itch | 5
  Erythema | 3
  Vertigo/dizziness | 44
  Cough/rhinitis/sore throat | 9
  Itchy | 9
  Drowsiness | 9
  Syncope/loss of consciousness | 18
  Hypesthesia/paresthesia | 7
  Chest pain/chest tightness | 8
  Stomach ache/dyspepsia | 6
  Dyspnea/tachypnea | 14
  Seizure | 3
  Paralysis/paresis | 3
  Slurred speech | 3
  Hyperhidrosis | 2
  Insomnia | 1

ADVERSE EVENTS:
Time Frame: The secondary data analysis of structured AE data conducted from 15-Mar-2023 to 03-Apr-2023(approximately 20 days) included AEs reported following administration of BNT162b2 mRNA SARS-CoV-2 vaccine from 21-Aug-2021 to 14-Dec-2022(approximately 1.3 years)
Description: This was a retrospective, observational study for secondary data collection and analysis of structured data regarding AEs reported in Indonesia NC AEFI database, following administration of BNT162b2 mRNA vaccine.
Arm/Group | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose
All-Cause Mortality (participants affected / at risk) | 3/150 | 2/110
Serious Adverse Events (participants affected / at risk) | 16/150 | 5/110
Other Adverse Events (participants affected / at risk) | 134/150 | 105/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose (N=150) | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose (N=110)
Cardiac arrest (Cardiac disorders) | 5 | 0
Ischemic stroke (Nervous system disorders) | 5 | 0
Hemorrhagic stroke (Nervous system disorders) | 2 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Diabetic ketoacidosis (Endocrine disorders) | 1 | 1
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abortus (Reproductive system and breast disorders) | 1 | 0
Hellp syndrome (Reproductive system and breast disorders) | 0 | 1
Caries dentist (Gastrointestinal disorders) | 1 | 0
Anaphylactic shock (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 mRNA SARS-CoV-2 Vaccine: Primary Dose (N=150) | BNT162b2 mRNA SARS-CoV-2 Vaccine: Booster Dose (N=110)
(General disorders) | 134 | 105 — AEs reported here are based on only sign and symptoms and were not investigated further (secondary data collection), hence diagnosis was unknown.

LIMITATIONS AND CAVEATS:
A total of 72,394,389 participants (48,425,165 [primary dose] and 23,969,029 [booster dose] received BNT162b2 mRNA SARS-CoV-2 vaccine. Adverse events were reported in 260 participants following administration of the BNT162b2 mRNA vaccine, starting from the time of vaccine availability in Indonesia and data was obtained for these 260 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT05621239/Prot_SAP_000.pdf